CLINICAL TRIAL: NCT05565378
Title: A Phase 2, Randomized, Open-label, Platform Study Utilizing a Master Protocol to Evaluate Novel Immunotherapy Combinations in Participants With Previously Untreated, Locally Advanced/Metastatic, Programmed Death Ligand 1-Selected Non-Small-Cell Lung Cancer
Brief Title: A Platform Study of Novel Immunotherapy Combinations in Participants With Previously Untreated, Advanced/Metastatic Non-Small-Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: iTeos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 213824; 2021-005115-32 (EudraCT Number); GALAXIES LUNG-201 (Other: Study Identifier)
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer, Non-Small Cell
Keywords: Belrestotug; Dostarlimab; EOS884448; GSK6097608; GSK4428859A; Nelistotug; Non-small-cell lung cancer; Pembrolizumab; Programmed death ligand 1; Programmed death protein 1 Inhibitor; Immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; dostarlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Pembrolizumab Monotherapy (Active Comparator): Participants will be administered with pembrolizumab as monotherapy in a fixed dose.
  Interventions: Drug: Pembrolizumab
- Dostarlimab Monotherapy (Experimental): Participants will be administered with dostarlimab as monotherapy in a fixed dose.
  Interventions: Drug: Dostarlimab
- Substudy 1A (Experimental): Participants will be administered with dostarlimab in a fixed dose followed by belrestotug in a fixed dose (Dose A).
  Interventions: Drug: Dostarlimab; Drug: Belrestotug
- Substudy 1B (Experimental): Participants will be administered with dostarlimab in a fixed dose followed by belrestotug in a fixed dose (Dose B).
  Interventions: Drug: Dostarlimab; Drug: Belrestotug
- Substudy 1C (Experimental): Participants will be administered with dostarlimab in a fixed dose followed by belrestotug in a fixed dose (Dose C).
  Interventions: Drug: Dostarlimab; Drug: Belrestotug
- Substudy 2A (Experimental): Participants will be administered with dostarlimab, fixed dose belrestotug, and fixed dose nelistotug
  Interventions: Drug: Dostarlimab; Drug: Belrestotug; Drug: Nelistotug

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab will be administered.
  Arms: Pembrolizumab Monotherapy
Drug: Dostarlimab — Dostarlimab will be administered
  Other Names: GSK4057190
  Arms: Dostarlimab Monotherapy; Substudy 1A; Substudy 1B; Substudy 1C; Substudy 2A
Drug: Belrestotug — Belrestotug will be administered.
  Other Names: EOS884448; GSK4428859A
  Arms: Substudy 1A; Substudy 1B; Substudy 1C; Substudy 2A
Drug: Nelistotug — Nelistotug will be administered.
  Other Names: GSK6097608
  Arms: Substudy 2A

SUMMARY:
This study will monitor the safety of novel immunotherapy combinations in participants with Programmed death ligand-1 (PD L-1) high (Tumor cells [TC]/ Tumor proportion score [TPS] >= 50%), previously untreated, unresectable, locally advanced or metastatic non-small cell lung cancer (NSCLC). Drug name mentioned as Belrestotug, GSK4428859A, and EOS884448 are all interchangeable for the same compound. In the rest of the document, the drug will be referred to as Belrestotug.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of locally advanced unresectable NSCLC not eligible for curative surgery and/or definitive radiotherapy with or without chemotherapy or metastatic NSCLC (squamous or non squamous)
* No prior systemic therapy for their locally advanced or metastatic NSCLC
* Provides a fresh tumor tissue sample or archival sample collected within 2 years prior to screening
* PD-L1-high (TC/TPS >= 50%) tumor
* Measurable disease based on RECIST 1.1, as determined by the investigator
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1
* Adequate Baseline organ function
* Female participants of childbearing potential must use adequate contraception

Exclusion Criteria:

* Has NSCLC with a tumor that harbors any of the following molecular alterations: EGFR and /or ALK translocations mutations that are sensitive to available targeted inhibitor therapy, Any other known genomic aberrations or oncogenic driver mutations for which a locally approved targeted therapy is available for first-line treatment of locally advanced or metastatic NSCLC.
* Had major surgery within 4 weeks or lung radiation of >30 Gy therapy within 6 months prior to the first dose of study intervention
* Received prior therapy with any immune checkpoint inhibitors
* Never smoked, defined as smoking <100 tobacco cigarettes in a lifetime
* Has an invasive malignancy or history of invasive malignancy other than the disease under study within the last 5 years (clinical exceptions apply as per protocol)
* Symptomatic, untreated, or actively progressing, brain metastases or any leptomeningeal disease (regardless of symptomatology, treatment status, or stability)
* Autoimmune disease or syndrome that required systemic treatment within the past 2 years
* Receiving systemic steroid therapy <= 3 days prior to first dose of study intervention or any form of immunosuppressive medication
* Received any live vaccine <= 30 days prior to first dose of study intervention
* Any history of idiopathic pulmonary fibrosis, organizing pneumonia, drug induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis
* History or evidence of cardiac abnormalities
* Current unstable liver or biliary disease
* Severe infection within 4 weeks prior to the first dose of study intervention
* Positive for tuberculosis, human immunodeficiency virus (HIV) infection, hepatitis B surface antigen, or hepatitis C
* Has advanced, symptomatic, or visceral spread and is considered to be at imminent risk of life-threatening complications (including, but not limited to, massive uncontrolled effusions [e.g., pleural, pericardial, peritoneal])
* Is currently participating in or has participated in a study of an investigational therapy within 4 weeks prior to the first dose of study intervention
* Has a history of allogeneic tissue/stem cell transplant or solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2027-02-26 (Estimated); Study Completion 2027-02-26 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Up to 228 weeks
Number of Participants with TEAEs or SAEs leading to dose modifications or treatment discontinuation | Up to 228 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (89):
- United States (4):
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Morgantown, West Virginia
- Argentina (7):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Cipoletti Rio Negro
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aire
  - GSK Investigational Site, Florida
  - GSK Investigational Site, Mar del Plata
  - GSK Investigational Site, San Juan
  - GSK Investigational Site, Santa Fe
- GSK Investigational Site, Wilrijk, Belgium
- Brazil (4):
  - GSK Investigational Site, Barretos
  - GSK Investigational Site, Porto Alegre
  - GSK Investigational Site, São Paulo
  - GSK Investigational Site, Vitória
- Finland (4):
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
  - GSK Investigational Site, Vaasa
- France (5):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Quimper
  - GSK Investigational Site, Strasbourg
- Germany (5):
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Essen
  - GSK Investigational Site, Großhansdorf
  - GSK Investigational Site, Heidelberg
  - GSK Investigational Site, Jena
- Greece (6):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Haidari - Athens
  - GSK Investigational Site, Larissa
  - GSK Investigational Site, PapagosAthens
  - GSK Investigational Site, Pylaia Thessaloniki
  - GSK Investigational Site, Thessaloniki
- Hungary (3):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Gyöngyös
  - GSK Investigational Site, Tatabánya
- Italy (5):
  - GSK Investigational Site, Avellino
  - GSK Investigational Site, Bergamo
  - GSK Investigational Site, Genova
  - GSK Investigational Site, Pisa
  - GSK Investigational Site, Verona
- Japan (6):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saitama
- Mexico (2):
  - GSK Investigational Site, Guadalajara
  - GSK Investigational Site, San Luis Potosí City
- Netherlands (4):
  - GSK Investigational Site, Enschede
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Leeuwarden
  - GSK Investigational Site, Utrecht
- Poland (3):
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Prabuty
  - GSK Investigational Site, Siedlce
- Portugal (4):
  - GSK Investigational Site, Gaia
  - GSK Investigational Site, Guimarães
  - GSK Investigational Site, Lisbon
  - GSK Investigational Site, Porto
- South Africa (2):
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Parktown
- South Korea (3):
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon Gyeonggi-do
- Spain (8):
  - GSK Investigational Site, Badajoz
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Las Palmas de Gran Canar
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, PamplonaNavarra
  - GSK Investigational Site, Valencia
- Thailand (5):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
  - GSK Investigational Site, Kho Hong Hat Yai
  - GSK Investigational Site, Khon Kaen
  - GSK Investigational Site, Pathum Thani
- Turkey (Türkiye) (4):
  - GSK Investigational Site, Samsun, Atakum
  - GSK Investigational Site, Ankara
  - GSK Investigational Site, Antalya
  - GSK Investigational Site, Istanbul
- GSK Investigational Site, Abu Dhabi, United Arab Emirates
- United Kingdom (3):
  - GSK Investigational Site, Middlesbrough
  - GSK Investigational Site, Middlesex
  - GSK Investigational Site, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/